CLINICAL TRIAL: NCT06660446
Title: Ejercicio Físico Durante El Tratamiento De Quimioterapia Como Programa Adyuvante En Pacientes Con Linfoma: Estudio EDONOLA
Brief Title: Exercise During Chemotherapy Treatment As Adjuvant Program in Patients with Lymphoma: EDONOLA Study.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biogipuzkoa Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EDONOLA
Record Dates: First submitted 2024-10-07; First posted 2024-10-28 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Lymphoma
Keywords: Lymphoma; Physical Exercise; Fatigue; Cardiorespiratory capacity; Life Quality
MeSH Terms: conditions — Lymphoma; Motor Activity; Fatigue | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): The control group will receive the usual care and indications.
- Intervention Group (Experimental): The interventional group will add a exercise program.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — The lymphoma unit of the Donostia University Hospital (HUD) is part of the Onkofrail project that analyzes the impact of a physical activity in older cancer patients. The Onkofrail study has included everything type of solid tumors and very diverse treatments, which is a limitation methodology that could condition the analysis of the results. Therefore, the need of proposing a new PE project in a homogeneous population such as that of people with lymphoma, the most prevalent hemopathy in our environment, which has a great survival, but present important adverse effects secondary to treatment systemic.
  Arms: Intervention Group

SUMMARY:
In people diagnosed with lymphoma receiving immunochemotherapy treatment, a combined exercise intervention, as opposed to the general recommendations, will achieve: 1.Improve cardiorespiratory fitness, strength, psychological well-being and quality of life. //2.Reduce fatigue//3.Reduce frailty

There is an association between some biological biomarkers with physical capacity and frailty.

DETAILED DESCRIPTION:
In this study, the effectiveness of an individualized adjuvant exercise program will be analyzed in a homogeneous population of people diagnosed with lymphoma in active treatment. Taking into account the limited scientific evidence that currently exists in people affected by lymphoma and active treatment, the study could be of great relevance when it comes to providing scientific evidence in this very little field studied. The study will try to respond to the evident need to focus the research area on supervised exercise in people with lymphoma in a way innovative, with the aim of generating new hypotheses that overcome existing limitations and facilitate the introduction of this type of interventions into the health system. The present study will also analyze the effect of exercise from a gender perspective, an aspect not systematically studied until now, providing a new vision on the baseline differences and after intervention of a program based on of sex.

The study will include adults with lymphoma with special focus on the subanalysis of the group of patients equal or more than 70 years old. The lymphoma unit of the Donostia University Hospital (HUD) is part of the Onkofrail project that analyzes the impact of a physical activity in older cancer patients. The Onkofrail study has included everything type of solid tumors and very diverse treatments, which is a limitation methodology that could condition the analysis of the results. Therefore, the need of proposing a new exercise project in a homogeneous population such as that of people with lymphoma, the most prevalent hemopathy in our environment, which has a great survival, but present important adverse effects secondary to treatment systemic. 30 people with lymphoma and treatment have been included in the Onkofrail study asset. The preliminary results of said pilot study have been used for the design of this new study, making adaptations, both in the recruitment time, as well as inclusion and exclusion criteria, which guarantee and optimize the correct research development.

Main objective:

The main objective is to assess whether a supervised (2 days/week) combined (resistance+aerobic interval training) exercise intervention, plus 2 days/week unsupervised for 20 weeks improves cardiorespiratory fitness (CRF) in people diagnosed with lymphoma undergoing chemotherapy, compared to a control group receiving only general recommendations.

Secondary objectives:

1. To estimate cardiorespiratory capacity (VO2peak) through a field test Modified Shuttle Walking Test (MSWT) and other covariates related to body composition, heart rate, among others. Validation of the predictive model.
2. To characterise and define the profile of the population diagnosed with lymphoma at the physical, emotional, and biochemical (biomarker) and immune system level prior to an intervention with exercise.
3. To investigate whether the implementation of an exercise programme adjuvant to immunochemotherapy treatment modifies fatigue, adherence (actual dose-intensity), and toxicity related to clinical treatment.
4. To analyse whether the intervention with exercise is effective in increasing strength levels, improving quality of life and sleep.
5. To clarify whether there are sex differences in the efficacy of the exercise programme adjuvant to immunochemotherapy treatment.
6. To analyse the benefit of adding exercise programmes in different subgroups of people with lymphoma, with a special focus on the group of patients aged ≥70 years, with the aim of maximising the cost-effectiveness of implementation in the care routine in all patients.
7. To analyse the degree of adherence to the programme: degree of attendance at planned sessions and percentage of participants who complete the post-intervention evaluation.
8. To report the degree of satisfaction by people affected by lymphoma, as reported in an interview.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years old.
* Diagnosis of lymphoma with histological confirmation and requirement of systemic treatment including chemotherapy.
* Time available (80 minutes, two days a week for 20 weeks) to carry out physical exercise sessions.
* Have a mobile phone to be able to contact the person and download the physical activity level app.
* Eastern Cooperative Oncology Group performance status (ECOG) ≤2.
* Life expectancy >12 months.
* Availability and desire to participate throughout the study period.

Exclusion Criteria:

* Have a contraindication to moderate-high intensity exercise.
* Other significant medical disorders: including psychiatric illnesses chronic or recurrent; intellectual disability, musculoskeletal problems, cardiac or pulmonary disorders that interfere with physical exercise; other malignant tumors in the last five years, with the exception of therapeutically controlled skin cancer; any other illness that may be seen affected or aggravated by physical exercise.
* Have plans to be outside city more than two weeks.
* People who are already physically active (that comply with the recommendations of WHO: > 150 minutes of exercise moderate/weekly, plus training force two days/week).
* Treatment based only with immunotherapy.
* Central nervous system involvement due to lymphoma.
* Have any important history that limit the capacity of the patient to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory fitness (CRF) | 20 weeks
  Measured by peak oxygen uptake (VO2peak) before starting chemotherapy treatment and after 20 weeks of intervention, using the cardiorespiratory exercise test.

SECONDARY OUTCOMES:
Sociodemographic, etiological and clinical health variables (A) | 20 weeks
  Recruitment Center (Donostia University Hospital, Galdakao University Hospital , Alava University Hospital)
Sociodemographic, etiological and clinical health variables (B) | 20 weeks
  Birthdate.
Sociodemographic, etiological and clinical health variables (C) | 20 weeks
  Biological sex (man, woman, I prefer not to answer)
Sociodemographic, etiological and clinical health variables (D) | 20 weeks
  Gender (man, woman, non-binary or I prefer not to answer)
Sociodemographic, etiological and clinical health variables (E) | 20 weeks
  Educational level (no studies, elementary, high school, vocational training, university, I prefer not to answer, others)
Sociodemographic, etiological and clinical health variables (F) | 20 weeks
  Home composition (single person, lives with couple, lives with family, institutionalized, I prefer not to answer, others)
Functionality and fragility variables at times T0, T1 and T2 (A.1.) | 20 weeks
  Muscle power and fragility --> SIT - TO STAND (STS) POWER: time to repeat the action 5 (sec)
Functionality and fragility variables at times T0, T1 and T2 (A.2.) | 20 weeks
  Muscle power and fragility --> FRAILTY TRAIT TEST SCALE (FTS-5): BMI (kg/m)2; running time (sec); grip strength (kg); Progressive Romberg Test (positive/negative).
Functionality and fragility variables at times T0, T1 and T2 (B.1.) | 20 weeks
  G8 Scale (0-17 pts)
Functionality and fragility variables at times T0, T1 and T2 (B.2.) | 20 weeks
  Fried Frailty Phenotype (0-5 pts)
Functionality and fragility variables at times T0, T1 and T2 (C) | 20 weeks
  Physical Condition: Modified Shuttle Walking Field Test (meters)
Functionality and fragility variables at times T0, T1 and T2 (D) | 20 weeks
  UPPER BODY MUSCLE STRENGTH (HANGRIP) (Newton)
Functionality and fragility variables at times T0, T1 and T2 (E) | 20 weeks
  Body composition --> Height (cm); Weight (kg); Waist circumference (cm); hip circumference (cm); body mass index (kg/m2); fat free mass (kg and %); fat mass (kg and %); total body water (kg and %); phase angle (º); systolic blood pressure (mmHG); diastolic blood presure (mmHg); resistance (Ω); reactance (Ω).
Functionality and fragility variables at times T0, T1 and T2 (F) | 20 weeks
  Physical activity level --> Global Questionnaire on Physical Activity (GPAQ)
Functionality and fragility variables at times T0, T1 and T2 (G) | 20 weeks
  Sleep Quality --> Epworth Sleepiness Scale (ESS EPWORTH) (0-24 pts)
Functionality and fragility variables at times T0, T1 and T2 (H) | 20 weeks
  Acelerometry (h/d)
Patient Reported Results (A) | 20 weeks
  Quality of Life Questionnaire --> Hematological Malignancy - Patient Reported Outcome (HM-PRO) at times T0, T1 and T2 (Nothing, mild and serious)
3. Patient-reported results (PRO): | 20 weeks
  EORTC QLQ - FA13
Biomarkers | 20 weeks
  Inflammation (pg/ml or ng/ml), Hematological (pg/ml or ng/ml), Endocrine Nutritional (pg/ml or ng/ml), Immunosenescence (pg/ml or ng/ml),
Variables of Geriatric Assessment (VGA) comprehensive in patients (A) | 20 weeks
  Gijon Scale (3-15 pts)
Variables of Geriatric Assessment (VGA) comprehensive in patients (B) | 20 weeks
  Basic Activity of Dialy Living (BADL) - Barthel Scale (0-10 pts)
Variables of Geriatric Assessment (VGA) comprehensive in patients (C) | 20 weeks
  Instrumental Activity of Dialy Livings (IADL) - Lawton Scale (0-8 pts)
Variables of Geriatric Assessment (VGA) comprehensive in patients (D) | 20 weeks
  Cognitive Function - Pfeiffer Test (0-10 pts)
Variables of Geriatric Assessment (VGA) comprehensive in patients (E) | 20 weeks
  Nutritional Status - Mini Nutritional Assessment Short-form (MNA.SFI) (0-14 pts)
Variables of Geriatric Assessment (VGA) comprehensive in patients (F) | 20 weeks
  Polypharmacy (number of chronica drug consumed by the participant)
Variables of Geriatric Assessment (VGA) comprehensive in patients (G) | 20 weeks
  Geriatric Syndromes - Immobility and pressure ulcers (Yes/No); instability and falls (Yes/No); urinary and faecal incontinence (Yes/No); dementia and acute confusional syndrome ( Yes//No); malnutrition (Yes/No); alterations in sight and hearing (Yes/No);constipation, faecal impaction (Yes/No);depression/insomnia (Yes/No)
Variables of Geriatric Assessment (VGA) comprehensive in patients (H) | 20 weeks
  Pain - Visual Analogue Scale (VAS) (0-10 pts)
Variables of Geriatric Assessment (VGA) comprehensive in patients (I) | 20 weeks
  Emotional Distress - Stress Thermometer (0-10 pts)
Treatment data and results after the intervention (T2) (A) | 20 weeks
  Treatment Suspension (Yes/No)
Treatment data and results after the intervention (T2) (B) | 20 weeks
  Dose Reduction (Yes/No)
Treatment data and results after the intervention (T2) (C) | 20 weeks
  Treatment percentage completed (%)
Treatment data and results after the intervention (T2) (D) | 20 weeks
  Treatment Completion (Yes/No)
Assessment of the intervention at T2 (A) | 20 weeks
  Adverse events associated with intervention (Number of adverse events)
Assessment of the intervention at T2 (B) | 20 weeks
  Satisfaction with the intervention (Yes/No)
Assessment of the intervention at T2 (C) | 20 weeks
  Adherence to the intervention (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Izaskun Zeberio Etxetxipia, Principal Investigator — Hospital Donostia
Locations (3):
- Spain (3):
  - Hospital Universitario Araba (HUA), Vitoria - Gateiz, Araba
  - Hospital Universitario Galdakao (HUG), Galdakao, Bizkaia
  - Hospital Universitario Donostia (HUD), San Sebastián, Guipuzcoa